CLINICAL TRIAL: NCT05022134
Title: A Prospective, Quasi-experimental Study to Evaluate the Feasibility of CHOICE-AYA for Unintended Pregnancy Prevention in Adolescents and Young Adults (AYA) Experiencing Homelessness.
Brief Title: Evaluating the Impact of CHOICE-AYA on Contraceptive Use, Continuation and Satisfaction
Acronym: CHOICE-AYA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Stephani Stancil, Assistant Professor, Department of Pediatrics, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00001846
Record Dates: First submitted 2021-08-09; First posted 2021-08-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Contraception Behavior; Sexual Behavior; Reproductive Behavior
Keywords: Adolescent; Contraception
MeSH Terms: conditions — Contraception Behavior; Sexual Behavior; Reproductive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (CHOICE-AYA) (Experimental): The impact of CHOICE-AYA contraceptive counseling on contraceptive use, satisfaction, and continuation will be assessed.
  Interventions: Behavioral: CHOICE-AYA

INTERVENTIONS:
Behavioral: CHOICE-AYA — Adapted contraceptive counseling specific to AYA experiencing homelessness

SUMMARY:
This is a prospective study involving two phases: 1) adaptation and 2) intervention, in adolescents aged 14-21 experiencing homelessness. The overarching goal is to develop and evaluate the effectiveness and feasibility of a counselling intervention to improve access to contraception among AYA experiencing homelessness. During the first phase, referred to as the adaption phase, we will rely on collective input from formative groups of AYA experiencing homelessness to adapt the CHOICE counselling intervention for this underserved and under-resourced population. In the second phase, referred to as the intervention phase, we will evaluate the effectiveness and feasibility of the adapted intervention (CHOICE-AYA).

DETAILED DESCRIPTION:
This study will adapt an evidence-based contraceptive counseling intervention (CHOICE) using input from the formative groups of AYA experiencing homelessness and study the impact of the adapted counseling (CHOICE-AYA) on contraceptive use, continuation, and satisfaction in a specialized community care setting. After informed consent is obtained, participants will receive the CHOICE-AYA counseling intervention by trained clinic staff. Provision of contraception based on participant choice will occur through the clinic provider same day.

Participants will be sent links to complete the follow-up surveys at 1, 3, 6, and 12 months. In addition, Clinic staff (e.g., prescribers and nurses) will be sent electronic surveys following randomly selected study visits.

Findings will inform best practices for this vulnerable population and provide foundational evidence for future studies focused on expanding care to other sites that serve this group.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults experiencing homelessness and housing instability (defined as those seeking care at our community-based clinic on the campus of a youth shelter) aged 14-21 who have female reproductive organs (In Missouri, youth aged ≤13 are not legally able to consent to sex)
* English speaking
* Prior sexual activity or anticipated future sexual activity that creates the risk of pregnancy
* Either not currently on hormonal contraception OR interested in switching methods

Exclusion Criteria:

* AYA currently seeking pregnancy in the next 3 months
* AYA with a severe developmental or cognitive delay that interferes with the ability to engage in consensual reproductive sex (determined by the investigator)

Ages: 14 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Contraceptive uptake | Study Day 1
  Rates of reliable contraceptive use

SECONDARY OUTCOMES:
Contraceptive satisfaction | 1, 3, 6, and 12 months post intervention
  brief likert-style survey assessing whether they are still on the method, how satisfied they are with this method
Contraceptive continuation | 1, 3, 6, and 12 months post intervention
  brief survey
Feasibility of intervention (perceived by clinic staff and participants) | Post-visit
  Brief survey based on Bowen's constructs of feasibility

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Research Institute, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No